CLINICAL TRIAL: NCT06108245
Title: The Impact of Values Clarification on Motivation to Declutter in People with Hoarding Problems: a Randomized Control Trial of a Prototype Mobile App Intervention
Brief Title: An Initial Test of Prototype Mobile App Interventions for Decluttering
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mississippi State University (Other)
Responsible Party: Principal Investigator, Jennifer Krafft, Assistant Professor, Mississippi State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-23-253
Record Dates: First submitted 2023-10-04; First posted 2023-10-30 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-11

CONDITIONS: Hoarding
Keywords: Clutter; Values Clarification; mHealth; Mobile app; Acceptance and Commitment Therapy
MeSH Terms: conditions — Hoarding; Speech Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned with equal likelihood to receive the values clarification prototype mobile application, the self-reflection prototype mobile application, or no treatment. After 8 weeks, participants who are in the no treatment group will be able to access both applications, and participants in either app group will be able to access the other app.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Values Clarification Condition (Experimental): Participants will be asked to respond to values clarification prompts twice a day over 28 days [4 weeks]. In each session, participants will receive a randomly assigned writing prompt from a pool of four categories: hierarchical, conditional, distinction, and perspective-taking prompts. In the initial session, participants will be asked to respond to a brief set of questions pertaining to their hoarding behavior in the past 12 hours and their motivation to declutter right now. From that point on, participants will respond to a brief set of questions before each writing prompt pertaining to their hoarding behaviors in the time since the previous writing prompt. After the writing prompt, they will be asked about how motivated they are to declutter right now. Each writing prompt is anticipated to take up to 10 minutes to complete and participants will receive notifications to use the app twice daily in addition email reminders twice a week to engage with the app.
  Interventions: Behavioral: Values Clarification Mobile Application
- Self-Reflection Condition (Placebo Comparator): Participants in this condition will be asked to respond to a set of randomly selected self-reflection prompts twice a day over 28 days [4 weeks]. As with the experimental condition, participants in the initial session will be asked to respond to a brief set of questions pertaining to their hoarding behavior in the past 12 hours and their motivation to declutter right now. From that point on, participants will be asked to respond to a brief set of questions before each writing prompt pertaining to their hoarding behaviors in the time since the previous writing prompt. After the writing prompt, they will be asked about how motivated they are to declutter right now. Each writing prompt is anticipated to take up to 10 minutes to complete, and participants will receive notifications to use the app twice daily in addition to email reminders twice a week to engage with the app.
  Interventions: Behavioral: Self-Reflection Mobile Application
- Waitlist Condition (No Intervention): Participants assigned to the waitlist will not receive access to any intervention for 8 weeks. After 8 weeks, they will receive access to either the values clarification or self-reflection mobile application.

INTERVENTIONS:
Behavioral: Values Clarification Mobile Application — Participants in the intervention group will be asked to answer a series of values clarification writing prompts twice a day over four weeks.
  Arms: Values Clarification Condition
Behavioral: Self-Reflection Mobile Application — Participants in the psychological placebo group will be administered writing prompts in the same format and frequency as the values intervention, but with prompts focused on self-reflection related to clutter and organization.
  Arms: Self-Reflection Condition

SUMMARY:
The aim of the study is to investigate whether values clarification writing prompts administered via a prototype mobile application can help enhance motivation and facilitate decluttering in individuals with hoarding problems. This randomized control trial will help to (1) assess whether values clarification can improve outcomes in hoarding treatment by increasing motivation, (2) clarify which specific values clarification procedures are most beneficial, and (3) evaluate the impact of values clarification on overall symptoms and well-being. Participants will be randomly assigned to either the experimental group (receiving the values clarification intervention), psychological placebo group (self-reflection intervention), or the no intervention waitlist group.

DETAILED DESCRIPTION:
This randomized control trial study aims to investigate the efficacy of a values clarification prototype mobile application intervention in enhancing motivation and facilitating decluttering in individuals with clinical levels of hoarding symptoms. Participants will be recruited using a variety of recruitment methods (e.g., Google Ads, posts on relevant online groups such as Facebook groups, posting flyers, and provider referrals). Interested participants will first complete a pre-screen asking about their age, country of residence, and whether they own an appropriate mobile device (i.e. iOS or Android). Eligible participants, who must be at least 18 years old and residing in the United States, will be provided with a consent form to sign and then directed to further screening to determine whether they meet the clinical cutoff for hoarding symptoms. Individuals who decline to participate or are screened as ineligible will be screened out and provided with a brief list of other resources they may access for clutter/hoarding problems. The researchers also reserve the right to screen individuals out if they are suspected to be bots or invalid participants. Individuals who consent and are screened as eligible will be redirected to complete a baseline survey and then randomly assigned to one of three groups with equal probability: (1) Experimental group with the values clarification mobile application, (2) psychological placebo group with the self-reflection mobile application, and (3) no-treatment waitlist group. Four weeks after baseline, participants will be asked to complete a post-treatment survey and eight weeks after baseline, participants will be asked to complete a final, follow-up survey. The no-treatment waitlist participants will be given the opportunity to download and use either prototype mobile app, and participants assigned to use one of the apps will be given the opportunity to use the alternative app.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older.
2. Living in the USA.
3. Owning an Android or iOS mobile device.
4. Meeting the clinical cutoff scores for the Saving Inventory-Revised and Clutter Image Rating scales.
5. Seeking help for clutter and/or hoarding.
6. Interested in testing a self-help prototype mobile app intervention.

Exclusion Criteria:

1. 17 years or younger.
2. Living outside the USA.
3. Not owning an Android or iOS mobile device.
4. Scoring below the clinical cutoff scores for the Saving Inventory-Revised and Clutter Image Rating scales.
5. Not seeking help for clutter and/or hoarding.
6. Not interested in testing a self-help prototype mobile app intervention.
7. Not having the fluency in English sufficient to understand study materials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
Saving Inventory - Revised (SI-R; Frost et al., 2004) | Baseline, Posttreatment (4 weeks after baseline) and Follow-up (8 weeks after baseline)
  A self-report measure of hoarding symptoms grouped into three factors: excessive acquisition, difficulty discarding, and clutter. The SI-R consists of 23 items that are rated on a scale from 0 (e.g., no distress) to 4 (e.g., extreme distress). Scores range from 0 to 92, with higher scores indicate greater endorsement of hoarding disorder symptoms.

SECONDARY OUTCOMES:
Sheehan Disability Scale (Sheehan, Harnett-Sheehan, & Raj, 1996) | Baseline, Posttreatment (4 weeks after baseline) and Follow-up (8 weeks after baseline)
  A self-report measure of functional impairment due to symptoms. It consists of 3 items rated on a scale from 0 (not at all) to 10 (extremely). Scores range from 0 to 30, with higher scores indicate greater impairment. This measure has been adapted to ask about disability related to hoarding.
Activities of Daily Living in Hoarding Scale (ADL-H; Frost et al., 2013) | Baseline, Posttreatment (4 weeks after baseline) and Follow-up (8 weeks after baseline)
  A self-report measure of activities impaired by hoarding disorder. The ADL-H consists of 15 items rated on a scale from 0 (can do it easily) to 5 (unable to do). A "not applicable" response option is also provided. Total scores range from a minimum of 0 to a maximum of 75, with higher scores indicating greater impairment.
Values Clarity Questionnaire (VCQ; McLoughlin et al., unpublished manuscript) | Baseline, Posttreatment (4 weeks after baseline) and Follow-up (8 weeks after baseline)
  A self-report scale that measures how well respondents understand and can articulate their values. The VCQ consists of 7 items rated on a scale from 1 (strongly disagree) to 5 (strongly agree). Total scores range from a minimum of 7 to a maximum of 35, with higher scores indicating higher levels of clarity, understanding, and articulation of one's own values.
Valuing Questionnaire (VQ; Smout et al., 2013) | Baseline, Posttreatment (4 weeks after baseline) and Follow-up (8 weeks after baseline)
  A self-report questionnaire that measures the extent to which one is living in accordance with their values. The VQ consists of 10 items rated on a scale from 0 (not at all true) to 6 (completely true). Total scores range from 0 to 60, with higher scores indicating greater valued living.
Acceptance and Action Questionnaire for Hoarding (AAQH; Krafft et al., 2019) | Baseline, Posttreatment (4 weeks after baseline) and Follow-up (8 weeks after baseline)
  A self-report measure of hoarding-related psychological inflexibility. The AAQH consists of 14 items rated on a scale from 1 (never true) to 7 (always true). Total scores range from 14 to 98, with higher scores indicating greater hoarding-related psychological inflexibility.
Depression, Anxiety, and Stress Scales (DASS-21; Henry & Crawford, 2005) | Baseline, Posttreatment (4 weeks after baseline) and Follow-up (8 weeks after baseline)
  A self-report measure of symptoms related to depression, anxiety, and stress. The DASS-21 consists of 21 items rated on a scale from 0 (did not apply to me at all) to 3 (applied to me very much, or most of the time). Total scores range from 0 to 63, with higher scores indicating greater endorsement of depression, anxiety, and stress related symptoms.
Satisfaction with Life Scale (SWLS; Diener et al., 1985) | Baseline, Posttreatment (4 weeks after baseline) and Follow-up (8 weeks after baseline)
  A self-report measure assessing one's satisfaction with their life as a whole. The SWLS consists of 5 items rated on a scale from 1 (strongly disagree) to 7 (strongly agree). Scores range from 5 to 35, with higher scores indicating greater life satisfaction.
Random responding question (used in e.g. Krafft & Levin, 2021) | Baseline, Posttreatment (4 weeks after baseline) and Follow-up (8 weeks after baseline)
  Participants will be asked to choose one of the following statements that best describe their participation in the survey, noting that their answer does not impact their participation in the study in any way: "I answered every question carefully and honestly" (1); "I answered most questions carefully and honestly" (2); "I randomly responded and/or did not respond honestly to about half of the questions"(3); "I randomly responded and/or did not respond honestly to most questions"(4); and "I randomly responded and/or did not respond honestly to any questions"(5). Participants who score a 4 or 5 will be screened out for random responding.
Treatment Evaluation Inventory-Short Form (TEI-SF; Kelley et al., 1989) | Posttreatment (4 weeks after baseline)
  A self-report measure of treatment acceptability. Only administered to the experimental and placebo conditions.The TEI-SF consists of 7 items rated from 1 (strongly disagree) to 5 (strongly agree). Scores range from 7 to 35, with higher scores indicating higher levels of endorsement for treatment acceptability.
System Usability Scale (SUS; Bangor et al., 2008) | Posttreatment (4 weeks after baseline)
  A self-report measure of usability of a technological system. The SUS consists of 10 items rated on a scale from 1 (strongly disagree) to 5 (strongly agree). Scores are summed and doubled such that they range from 0 to 100 (as per the official scoring instructions), with high scores indicated greater usability. Only administered to the experimental and placebo conditions.
Credibility/Expectancy Questionnaire (CEQ; Devilly & Borkovec, 2000) | After using first website session (approximately 0-1 weeks after baseline)
  A self-report measure of the perceived credibility of and expectations toward a treatment. Only administered to the experimental and placebo conditions. The CEQ consists of 6 items, 3 for Credibility and 3 for Expectancy. An average score ranging from 1 to 9 will be calculated for Credibility, with higher scores a greater perception of the intervention's credibility by the participants. For the expectancy component, an average percentage score will be calculated ranging from 0% to 100%, with higher percentages indicating more positive expectations towards the treatment.
Novel satisfaction item 1 | Posttreatment (4 weeks after baseline)
  Participants will be asked an open-ended question to gather qualitative feedback on the intervention. Only assigned to the experimental and placebo conditions. The question is, "What did you like best about the prototype mobile app?"
Novel satisfaction item 2 | Posttreatment (4 weeks after baseline)
  Participants will be asked an open-ended question to gather qualitative feedback on the intervention. Only administered to the experimental and placebo conditions. The question is, "What was the most important thing you learned from the mobile app?"
Novel satisfaction item 3 | Posttreatment (4 weeks after baseline)
  Participants will be asked an open-ended question to gather qualitative feedback on the intervention. Only assigned to the experimental and placebo conditions. The question is, "What did you like least about the mobile app? Why did you like this the least?"
Novel satisfaction item 4 | Posttreatment (4 weeks after baseline)
  Participants will be asked an open-ended question to gather qualitative feedback on the intervention. Only assigned to the experimental and placebo conditions. The question is, "Do you have any other comments or suggestions regarding the mobile app?"

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Krafft, PhD, Principal Investigator — Mississippi State University
Locations (1):
- Mindfulness and Acceptance Processes Lab, Starkville, Mississippi, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to share fully deidentified data sets. We will remove any potentially identifying information including unusual demographics or combinations of demographics removed, but all other variables will be available to other researchers, journals or officials on reasonable request.
Supporting Information: Study Protocol
Time Frame: Within one year of the end of data collection, and remaining available indefinitely
Access Criteria: There are no specific access criteria. The request must have a valid research-related purpose.

REFERENCES:
- [Background] Brooke, J. (1996). SUS: A "quick and dirty" usability scale. In P. W. Jordan, B. Thomas, B. A. Weerdmeester, & I. L. McClelland (Eds.), Usability evaluation in industry (pp. 189-194). Taylor & Francis.
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119
- [Background] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493
- [Background] Frost RO, Hristova V, Steketee G, Tolin DF. Activities of Daily Living Scale in Hoarding Disorder. J Obsessive Compuls Relat Disord. 2013 Apr 1;2(2):85-90. doi: 10.1016/j.jocrd.2012.12.004. Epub 2012 Dec 25. PMID 23482436
- [Background] Frost RO, Steketee G, Grisham J. Measurement of compulsive hoarding: saving inventory-revised. Behav Res Ther. 2004 Oct;42(10):1163-82. doi: 10.1016/j.brat.2003.07.006. PMID 15350856
- [Background] Frost, R. O., Steketee, G., Tolin, D. F., & Renaud, S. (2008). Development and validation of the clutter image rating. Journal of Psychopathology and Behavioral Assessment, 30, 193-203.
- [Background] Henry JD, Crawford JR. The short-form version of the Depression Anxiety Stress Scales (DASS-21): construct validity and normative data in a large non-clinical sample. Br J Clin Psychol. 2005 Jun;44(Pt 2):227-39. doi: 10.1348/014466505X29657. PMID 16004657
- [Background] Kelley, M. L., Heffer, R. W., Gresham, F. M., & Elliott, S. N. (1989). Development of a modified treatment evaluation inventory. Journal of psychopathology and behavioral assessment, 11, 235-247.
- [Background] Bangor, A., Kortum, P. T., & Miller, J. T. (2008). An empirical evaluation of the system usability scale. Intl. Journal of Human-Computer Interaction, 24(6), 574-594.
- [Background] Krafft, J., & Levin, M. E. (2021). Does the Cognitive Fusion Questionnaire measure more than frequency of negative thoughts?. Journal of Contextual Behavioral Science, 22, 63-67.
- [Background] Krafft, J., Ong, C. W., Twohig, M. P., & Levin, M. E. (2019). Assessing psychological inflexibility in hoarding: The Acceptance and Action Questionnaire for Hoarding (AAQH). Journal of Contextual Behavioral Science, 12, 234-242.
- [Background] McLoughlin, S., Stapleton, A., & Hochard, K. D. (2022). Development and preliminary validation of the Value Clarity Questionnaire. PsyArXiv. https://doi.org/10.31234/osf.io/u97q3
- [Background] Sheehan DV, Harnett-Sheehan K, Raj BA. The measurement of disability. Int Clin Psychopharmacol. 1996 Jun;11 Suppl 3:89-95. doi: 10.1097/00004850-199606003-00015. PMID 8923116
- [Background] Smout, M., Davies, M., Burns, N., & Christie, A. (2014). Development of the valuing questionnaire (VQ). Journal of Contextual Behavioral Science, 3(3), 164-172.